CLINICAL TRIAL: NCT06939179
Title: Evaluation of the Effect of Face Mask Therapy and RPE Application on Blood Oxygen Levels
Brief Title: Effect of Face Mask Therapy on Blood Oxygen Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Burak Aydin, investigator, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-KAEK-77-23-04
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2023-12

CONDITIONS: Control Patients; Class III Malocclusion
Keywords: face mask therapy; rapid maxillary expansion; orthodontics
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: In our study, cases were divided into two test groups and one control group. One group will be administered a rapid upper jaw expansion protocol with a face mask device and will be asked questions about the airway and its quality. The rapid maxillary expansion appliance applied to this group is bonded hyrax type. In the other test group, a bonded appliance without an expansion effect on the upper jaw was designed and applied. A petit-type facemask appliance will be applied with the appliance and respiratory quality will be questioned.The control group was asked about their respiratory tract and quality on the day they were first admitted to our clinic, pulse oximetry measurements will be made and they were called back at the end of 6 months, which is the average face mask treatment period, and this process was repeated.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- non treated control group (Active Comparator): The control group was asked about their respiratory tract and quality on the day they were first admitted to our clinic, pulse oximetry measurements will be made and they were called back at the end of 6 months, which is the average face mask treatment period, and this process was repeated.
  Interventions: Other: Class III Malocclusion
- face mask with rapid maxillary expansion treated group (Experimental): group will be administered a rapid upper jaw expansion protocol with a face mask device and will be asked questions about the airway and its quality. The rapid maxillary expansion appliance applied to this group is bonded hyrax type.
  Interventions: Other: Class III Malocclusion
- face mask without rapid maxillary expansion group (Experimental): Thisgroup, a bonded appliance without an expansion effect on the upper jaw was designed and applied. A petit-type facemask appliance will be applied with the appliance and respiratory quality will be questioned.
  Interventions: Other: Class III Malocclusion

INTERVENTIONS:
Other: Class III Malocclusion — Class III malocclusion treatment
  Arms: face mask with rapid maxillary expansion treated group; face mask without rapid maxillary expansion group
Other: Class III Malocclusion — non treated Class III malocclusion
  Arms: non treated control group

SUMMARY:
Skeletal Class III malocclusions are characterized by maxillary retrusion, mandibular protrusion, or a combination of both. In growing individuals presenting with maxillary deficiency, the face mask appliance is widely recognized as one of the most effective and frequently utilized orthopedic interventions. The primary objective of face mask therapy is to stimulate forward and downward growth of the maxilla by disarticulating and activating the circummaxillary sutural system. The application of protraction forces via a face mask results in anterior displacement of the maxillary dentition, accompanied by lingual inclination of the mandibular incisors. Orthopedic effects of the appliance typically include forward and downward movement of the maxilla with a slight degree of upward rotation, posterior dental extrusion, and backward rotation of the mandible. Numerous studies have demonstrated that combining rapid maxillary expansion (RME) with face mask therapy enhances skeletal outcomes, especially when initiated during the early stages of growth. Delayed intervention is often associated with reduced orthopedic responsiveness.

Foersch et al. evaluated the effects of pre-treatment rapid maxillary expansion on face mask therapy outcomes and concluded that expansion positively influences sagittal skeletal changes. In the absence of expansion, greater dental compensation was observed, particularly in the transverse dimension. From a clinical standpoint, anterior crossbite correction can typically be achieved within approximately 3 to 4 months, depending on the severity of the malocclusion. However, establishing a stable overbite and molar relationship usually requires an additional 4 to 6 months of treatment. A prospective clinical study analyzing treatment outcomes in Class III patients reported that overjet correction occurred through 31% maxillary advancement, 21% mandibular retraction, 28% labial proclination of the maxillary incisors, and 20% lingual retroclination of the mandibular incisors. To compensate for potential adverse effects of late mandibular growth, overcorrection of the overjet and molar relationship has been recommended. RME has also been associated with significant anatomical and functional changes in the upper airway. Specifically, an increase in the width of the nasal cavity base leads to a reduction in nasal airway resistance and improvement in nasal respiration. Recent investigations have documented post-treatment increases in pharyngeal airway dimensions and corresponding enhancements in nasal breathing. In a clinical study involving 25 patients with Class III malocclusion due to maxillary deficiency, face mask therapy resulted in a significant increase in nasopharyngeal airway space, which remained stable after a four-year follow-up period. Another study comparing 18 patients treated with RME and face mask therapy against an untreated control group of 163 individuals demonstrated a statistically significant enlargement of the nasopharyngeal space in the treated group. Pulse oximetry operates based on two fundamental physical principles. First, arterial blood generates a pulsatile signal, while non-pulsatile signals originate from venous and capillary beds. Second, modern oximeters utilize light-emitting diodes (LEDs) emitting at wavelengths of 660 nm (red) and 940 nm (infrared), as oxyhemoglobin and deoxygenated hemoglobin display distinct absorption spectra at these wavelengths. In a study conducted by Niaki et al., among patients exhibiting mouth breathing patterns, 65.4% were classified as hypoxemic, while 34.6% had normal oxygen saturation levels. Gender analysis revealed that 31.4% of males and 40% of females demonstrated normal oxygen saturation.Mouth breathing has been shown to influence craniofacial growth and may contribute to the development of various malocclusion patterns. Conversely, specific malocclusion types can exacerbate oral breathing tendencies. It is important to acknowledge that oral respiration has a measurable impact on blood oxygen levels and overall respiratory function.

ELIGIBILITY:
Inclusion Criteria:

6-10 years of age Class III Malocclusion

-

Exclusion Criteria:

* +10 years of age

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
examination of oxygen level of Class III malocclusion | up to 6 months
  examination of oxygen levels with or without Class III Malocclusion treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided